CLINICAL TRIAL: NCT00996411
Title: Human Psychopharmacology of Salvinorin A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Roland Griffiths, Professor, Department of Psychiatry,, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: NA_00009081
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Healthy volunteers are being studied to evaluate the subject-rated, behavioral, and abuse liability effects of salvinorin A
MeSH Terms: conditions — Behavior | interventions — salvinorin A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- Salvinorin A (Experimental)
  Interventions: Drug: Salvinorin A

INTERVENTIONS:
Drug: Salvinorin A — This is an initial dose ranging study

SUMMARY:
This study is characterizing the subject-rated and behavioral effects of salvinorin A in healthy volunteers. The investigators hypothesize the salvinorin A will have hallucinogen-like effects.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Have a high school level of education
* Have a self-reported interest in spirituality and altered states of consciousness
* Have used hallucinogens (e.g., LSD, psilocybin mushrooms, Salvia divinorum) including having used Salvia divinorum or salvinorin A by the inhalation route (i.e., volunteers without histories of Salvia divinorum or salvinorin A use by the inhalation route will be excluded)
* Be 21 to 65 years old
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the volunteer does not routinely consume caffeinated beverages, he or she must agree not to do so on session days.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, within 24 hours of each drug administration. As described elsewhere, exceptions include daily use of caffeine.
* Be healthy as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocarroutine medical blood and urinalysis laboratory tests.

Exclusion Criteria:

General Medical Exclusion Criteria

* Cardiovascular conditions: uncontrolled hypertension, angina, a clinically significant ECG abnormality (e.g. atrial fibrillation), TIA in the last 6 months stroke, peripheral or pulmonary vascular disease
* Epilepsy with history of seizures
* Diabetes mellitus
* Females who are pregnant (positive pregnancy test) or nursing, or are not practicing an effective means of birth control
* Currently taking psychoactive prescription medication on a regular basis
* More than 20% outside the upper or lower range of ideal body weight according to Metropolitan Life height and weight table

Psychiatric Exclusion Criteria

* Current or past history of meeting DSM-IV criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I or II Disorder.
* Current severe Obsessive-Compulsive Disorder, Dysthymic Disorder, or Panic Disorder.
* Current or past history within the last 5 years of meeting DSM-IV criteria for alcohol or drug dependence (excluding caffeine and nicotine) or severe major depression.
* Have a first or second degree relative with schizophrenia, psychotic disorder (unless substance induced or due to a medical condition), or bipolar I or II disorder.
* Currently meets DSM-IV criteria for Dissociative Disorder, Anorexia Nervosa, Bulimia Nervosa, or other psychiatric conditions judged to be incompatible with establishment of rapport or safe exposure to salvinorin A.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2008-11; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Hallucinogen Rating Scale | Approximately 1 hour after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Roland Griffiths, Ph.D., Principal Investigator — Johns Hopkins University; Matthew W Johnson, Ph.D., Study Director — Johns Hopkins University
Locations (2):
- United States (2):
  - Behavioral Pharmacology Research Unit, Johnson Hopkins Univ. School of Med., Baltimore, Maryland
  - Behavioral Pharmacology Research Unit, Baltimore, Maryland